CLINICAL TRIAL: NCT05362617
Title: mFOLXOX6 Versus FOLFIRI for Colorectal Patients Recurrence After Oxaplatin Based Adjuvant Chemotherapy（NEW RECHALLENGE）- A Multicenter Open Prospective Randomized Controlled Trial
Brief Title: mFOLXOX6 Versus FOLFIRI for Colorectal Patients Recurrence After Oxaplatin Based Adjuvant Chemotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRE202001
Record Dates: First submitted 2021-08-15; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2021-08

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic colorectal cancer; Completion of adjuvant therapy; First line chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FOLFIRI (Experimental): Irinotecan 180 mg/m2 I.V 30-90 min，D1；
  LV 400 mg/m2 I.V.，D1；
  5-FU 400 mg/m2 IVP，d1,1200 mg/m2/d×2 days（Total:2400 mg/m2，Continuous intravenous infusion,46~48 hours,）
  Repeat Every 14 days
  Interventions: Drug: FOLFIRI
- mFOLFOX6 (Active Comparator): Oxaplatin 85 mg/m2 I.V 120 min，D1；
  LV 400 mg/m2 I.V.，D1；
  5-FU 400 mg/m2 IVP，d1,1200 mg/m2/d×2 days（Total:2400 mg/m2，Continuous intravenous infusion,46~48 hours,）
  Repeat Every 14 days
  Interventions: Drug: FOLFIRI

INTERVENTIONS:
Drug: FOLFIRI — FOLFIRI as first line chemotherapy versus mFOLFOX6 after adjuvant chemotherapy

SUMMARY:
A multicenter,open,prospective randomized controlled trial;11 study center in China; Plan to enroll 328 patients（ Power Analysis and Sample Size ）.Comparing FOLFIRI with mFOLFOX6,Superiority design.Investigate difference PFS,ORR,R0 resection rate,OS ,QoL and Safety from two regimens Stratification factors : Analyzing patients recurrence within 6-12months,and 12-18months .Obtain definite chemotherapy regimen shift opportunity for patients recurrence/metastasis after adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

18-75 years，male or female Colorectal adenocarcinoma Accepting more than 4 cycles oxaplatin based adjuvant chemotherapy after radical operation Reccurrence in 6-18 months after adjuvant chemotherapy At least one assessable lesions No intestinal obstruction ECOG 0-1 Estimated survival≥ 3 months CBC：WBC>4×109/L，PLT>80×109/L，Hb>90g/L， Liver function：ALT or AST < 2× normal maximum value， T-bile<1.5× normal maximum value without hepatic metastatic， ALT or AST < 5× normal maximum value， T-bile<1.5× normal maximum value with hepatic metastatic Cr<1.8mg/dl Signed informed consent

Exclusion Criteria:

Locally resectable lesions Grade 2-4 oxaliplatin induced neurotoxicity Arrhythmias，coronary heart disease，or congestive heart failure（NYHA≥grade 2） requiring treatment Poorly controlled hypertension HIV infected or active HBV or HCV infected Active serious infection Cachexia or organ function decompensation Multiple primary carcinoma except carcinoma in situ of skin and cervix Participate in other clinical studies at the same time Serious heart or brain disease Drug abuse or other serious psychosocial diseases Suspected trial drug allergy Other factors affecting patient safety and compliance Pregnant or lactating women，or fertility without adequate contraceptive measures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR（objective response rate） | At the end of Cycle 3（6 weeks after first chemotherapy）
  imaging evaluation

SECONDARY OUTCOMES:
PFS | At the end of Cycle 6(each cycle is 14 days)
  imaging evaluation PD
OS | At the end of Cycle 12(each cycle is 14 days)
  patient death
R0 resection rate R0 resection rate R0 resection rate R0 resection rate R0 resection rate | At the end of Cycle 12(each cycle is 14 days)
  sugery
QoL（quality of life） | At the end of Cycle 12
  Life state

CONTACTS AND LOCATIONS:
Locations (1):
- SAHZU, Hangzhou, Zhejinag, China

IPD SHARING:
Plan to Share IPD: No